CLINICAL TRIAL: NCT04969809
Title: Comparison of Atherogenic Risk Factors and Efficacy of Nutritional Treatment Among Adult Phenylketonuria Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Ajda Mezek, mag.diet., University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMezek
Record Dates: First submitted 2021-06-21; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Phenylketonurias; Nutritional and Metabolic Diseases
Keywords: adult phenylketonuria; nutrition therapy; cardiovascular diseases; nutrition and metabolic diseases
MeSH Terms: conditions — Phenylketonurias; Nutritional and Metabolic Diseases; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: We will invite approximately 50 adult patients with PKU who were or are still being managed in the PPB clinic of the Pediatric Clinic of the University Medical Center Ljubljana. It is estimated that half of the patients still fully or at least partially follow the dietary treatment, while half have abandoned the treatment and mostly no longer come for outpatient examinations.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients on diet (Experimental): We will invite approximately 50 adult patients with PKU who were or are still being managed in the PPB clinic of the Pediatric Clinic of the University Medical Center Ljubljana. It is estimated that half of the patients still fully or at least partially follow the dietary treatment.
  Interventions: Diagnostic Test: Ultrasound of the jugular veins; Dietary Supplement: addition of phenylalanine-free protein substitutes
- patients without diet (Experimental): Half of the patients have abandoned the diet treatment and mostly no longer come for outpatient examinations.
  Interventions: Diagnostic Test: Ultrasound of the jugular veins; Dietary Supplement: addition of phenylalanine-free protein substitutes

INTERVENTIONS:
Diagnostic Test: Ultrasound of the jugular veins — Ultrasound of the jugular veins to assess the thickness of the carotid intima media
Dietary Supplement: addition of phenylalanine-free protein substitutes — addition of phenylalanine-free protein substitutes for sufficient daily intake of essential amino acids and other vitamins and minerals and nutritional plan

SUMMARY:
Phenylketonuria is a rare metabolic disease that results from the absence or near-absence activity of the enzyme phenylalanine hydroxylase, which metabolizes the amino acid phenylalanine to tyrosine in the body. Accumulation of phenylalanine in the brain causes brain damage that leads to mental retardation, neurological complications, and movement disorders.

The study is inherited autosomal recessively. The basis of treatment is a low-protein diet with dietary supplements of aminoxlin without phenylalanine and with appropriate substitutes for micro and macronutrients needed for different ages. A low-protein diet regulates the level of phenylalanine in the blood. This is especially important in childhood.

In the study, which will basically consist of theoretical, experimental and numerical work, the investigators will limit to a specific population, i.e. to adult patients with phenylketonuria. The research is intended to prove the hypothesis that with proper nutritional treatment of phenylketonuria in adulthood, we can have a positive effect on the patient's well-being, better blood results and improved lifestyle.

The investigators intend to test this hypothesis by implementing a complex, multidisciplinary project that will include a comprehensive treatment of adult PKU patients. This will be based on a multidisciplinary approach with the inclusion of medical and nutritional treatment. As part of the project, the investigators, among other things, create questionnaires and analyze food diaries related to the mentioned areas.

Using various statistical techniques, the investigators analyze the impact of individual factors on the success of achieving the objectives of the proposed study. The original contribution to science will be the nutritional treatment of adult patients with phenylketonuria in Slovenia and the consequent reduction of health complications in adulthood of patients with phenylketonuria.

DETAILED DESCRIPTION:
Selection and presentation of the problem and formulation of goals Phenylketonuria (PKU) oz. Hyperphenylalaninemia (HPA) is a rare congenital metabolic disease (PPB) due to a lack of phenylalanine hydroxylase (PH) activity, which metabolizes the amino acid phenylalanine (Phe) to tyrosine in the body. The cause is a disease change in the PAH gene that encodes the enzyme PH. A baby is born healthy, but elevated Phe levels without proper treatment cause central nervous system damage and permanent mental retardation in the first months after birth. The disease is the first PPB to be detected by medicine with neonatal screening tests and also successfully treated with dietary treatment that excludes foods with a higher Phe content from the diet. In Slovenia, the screening test was introduced in 1979 and with a calculated incidence of PKU 1/6769 in Slovenia (Šmon et al., 2015), there are approximately 150 patients with PKU in the Slovenian registry, of which more than half are over 18 years of age.

Nutritional treatment is an important part of PKU treatment and should be performed for life according to modern guidelines (Cazzorla et al., 2018).

Dietary treatment of PKU is one of the strictest diets, where almost all foods containing protein are excluded from the food, ie all diets of animal origin (meat, milk and all dairy products, eggs) as well as all cereals, legumes and nuts. Patients consume only limited amounts of fruits and vegetables and special products with a removed protein content. They compensate for the protein deficiency with special Phe-free protein substitutes. Adult patients with PKU often do not reach the recommended levels of Phe in the blood (Green et al., 2019), as the consequences of abandoning the diet in adulthood are not as obvious and disturbing. By abandoning the diet, however, they also abandon follow-up in a specialist PPB clinic, and according to studies, more than 70% of adult patients with PKU (study in America) are no longer managed in metabolic clinics (Berry et al., 2013).

Successful disease management often requires a lifelong diet that provides an appropriately limited daily intake of Phe for growth and body regeneration with a small portion of essential amino acids, vitamins, and natural food elements, and the remaining missing portion of these dietary sources is added in the form of protein-fortified protein. , which does not contain the amino acid Phe (MacLeod et al., 2009). Phe tolerance (mg Phe / kg body weight / day) is the amount of Phe that PKU patients can consume daily while maintaining recommended blood Phe levels. An individual assessment is required due to the very diverse level of Phe hydroxylase enzyme activity still present (MacLeod et al., 2009). The measure of dietary success is an adequate value of serum Phe and the latest European recommendations in adulthood are between 120 - 600 μmol / L (van Spronsen et al., 2017; van Wegberg et al., 2017).

Research in recent years has shown significantly higher morbidity and health risk in adult patients with PKU. Part of the health problems are also more present in patients who continue dietary treatment, and there are even more problems in untreated patients (Burton et al., 2018).

Increased health risks have already been described, including the following medical conditions:

* Increased cardiovascular risk and increased atherogenic indicators (Azabdaftari et al., 2019)
* Higher body mass index (Robertson et al., 2013)
* The impact of disease and diet on bone density (Hansen et al., 2014)
* Nutritional deficits (Okano et al., 2016, Moseley et al., 2002)
* Higher proportion of brain dysfunction (Hoedt et al., 2012)
* Gastrointestinal dysbiosis (Verduci et al., 2020)
* Increased general comorbidity (Burton et al., 2018)

All these increased risks mean that this group of patients needs regular medical monitoring even in adulthood. It is known that a proportion of patients relax their diet and thus their Phe intake, but maintain a self-limiting diet with a low protein intake while not consuming a protein substitute (Das et al., 2014). Adequate daily protein intake is important as it ensures proper body protein synthesis and prevents catabolism (MacLeod et al., 2009).

The purpose of the research

Primary goal:

1. Use a questionnaire in patients to assess the differences between the group of patients on dietary treatment and the group of patients who discontinued treatment: demographic characteristics (gender, age, education, source of income, marital status), comorbidities or treatments, smoking , sleep disorders, self - assessment of physical activity, self - assessment of health.
2. To determine the effectiveness of the dietary intervention of individual nutrition counseling for reduced Phe intake in the blood and the balance of nutrients and elements in the diet by assessing the following indicators, before and after 6 months of intervention:

   * quantitative reduction of Phe consumption in the diet and adequacy of Phe amino acid preparation with the addition of vitamins and elements, which will be assessed by measurements in the blood: Phe, amino acids, vitamins, trace elements, methylmalonic acid in urine
   * Compliance assessment with analysis of food diaries (at the first examination and after 6 months)

Secondary objectives are:

1. Comparison of assessment of risk factors for atherogenesis between patients considering dietary treatment and among patients without dietary treatment with ultrasound of the jugular veins to assess the thickness of the carotid intima media and assessment of oxidative stress in the urine sample and body composition at the start of the study
2. Assessment of risk factors for atherogenesis before and after dietary intervention

   * Determine the change in body mass index, waist circumference before and after the intervention, blood pressure
   * Identify the change of selected laboratory atherogenic biomarkers (total lipidogram, Lp (a), homocysteine, CRP low, Il-6, TNF alpha, blood sugar, insulin) Presentation of methods

The investigators will invite approximately 50 adult patients with PKU who were or are still being managed in the PPB clinic of the Pediatric Clinic of the University Medical Center Ljubljana. It is estimated that half of the patients still fully or at least partially follow the dietary treatment, while half have abandoned the treatment and mostly no longer come for outpatient examinations.

The research will be conducted prospectively. Institution where the research will be conducted: Clinical Department of Endocrinology, Diabetes and Metabolic Diseases, Pediatric Clinic, University Medical Center Ljubljana, Bohoričeva 20, 1000 Ljubljana

Nutritional analyzes and interventional dietary counseling will be performed simultaneously with the regular medical control outpatient examination before the nutritional intervention and the analysis will be repeated after 6 months.

INTRODUCTORY REVIEW:

Ultrasound of the jugular veins to assess the thickness of the carotid intima media as a non-invasive biomarker of atherosclerosis (cIMT) will be performed by a specialist as a regular existing examination method during outpatient examination of the patient (non-invasive ultrasound probe MyLab Gamma with QIMT® software according to the manufacturer's instructions).

The first inspection will also include:

* Completion of a questionnaire (Physical Activity Questionnaire (International Physical Activity Questionnaire), Sleep Questionnaire (Insomnia Severity Questionnaire (ISI)),
* performing anthropometric measurements (body weight (kg), body height (cm), waist circumference (cm)) (validated scales, stadiometer, prescribed waist circumference measurement procedure)
* measurement of systolic and diastolic blood pressure (mmHg) and resting pulse,
* nutrition analysis (by completing nutrition diaries and / or an interview at the examination)
* taking a blood sample
* taking a urine sample
* body composition measurement - BIA
* OGTT testing

Nutrition analysis and interventional nutrition counseling will include:

Definition of diet To define the diet (energy and nutrient intake), the investigators use the diet diary (PD) of the patient's diet for three days (3 x 24 hours (I .: 0 months = before the 1st examination; PD 0)) and 3 x 24 hours, where patients food diary will be carefully reviewed by a dietitian and will be entered into the Prodi® program for further processing and calculation of detailed energy and nutrient intake. preparation of menus, composition of individual recipes and calculation of nutrient and energy intake.

Subjects will receive one hour of nutritional counseling in a diet counseling center by a clinical dietitian.

Nutritional counseling will be based on the nutritional assessment of the patient's condition and the direction of improvement - the development of a diet plan. The dietitian will make a motivational phone call each month. Written instructions will be given to the examinees.

REVIEW AFTER 6 MONTHS:

The inspection will include:

* filling in the sleep disorder questionnaire, self-assessment of physical activity, self-assessment of health
* performing anthropometric measurements (body weight (kg), body height (cm), waist circumference (cm)) (use of a validated balance, stadiometer, prescribed waist circumference measurement procedure)
* measurement of systolic and diastolic blood pressure (mmHg),
* nutrition analysis (by completing nutrition diaries and screening interviews)
* taking a blood sample
* taking a urine sample
* body measurement

ELIGIBILITY:
Inclusion Criteria:

* The study will include subjects over the age of 18 who have PKU or hyperphenylalaninemia and are expected to have dietary treatment according to expert recommendations. A prerequisite for entering the investigation will be a signed consent to participate in the investigation and the ability of the participant to have a good understanding of the content of the research and to fully participate in the interventional dietary process.

Exclusion Criteria:

* The investigators will not include adult patients who do not manage their diet on their own and need caregivers due to limited cognitive abilities (patients with late-diagnosed disease and neurological consequences of the disease) or who do not want to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
assess the differences between the group of patients with questionnaire | up to 6 months
  Use a questionnaire in patients to assess the differences between the group of patients on dietary treatment and the group of patients who discontinued treatment: demographic characteristics (gender, age, education, source of income, marital status), comorbidities or treatments, smoking , sleep disorders, self - assessment of physical activity, self - assessment of health.
Determination of the effectiveness of the dietary intervention of individual nutrition counseling for reduced Phe intake in the blood and the balance of nutrients and elements in the diet | up to 6 months
  Phe intake in the blood (µmol/L)

SECONDARY OUTCOMES:
Comparison of the assessment of risk factors for atherogenesis | 1 day
  ultrasound of the jugular veins to assess the thickness of the carotid intima media (percent)
Assessment of risk factors for atherogenesis before and after dietary intervention 1 | up to 6 months
  Determine the change in body mass index (kg/m²)
Assessment of risk factors for atherogenesis before and after dietary intervention 2 | up to 6 months
  waist circumference (cm)
Assessment of risk factors for atherogenesis before and after dietary intervention 3 | up to 6 months
  blood pressure (mm Hg)
Bioelectrical impedance analysis (BIA) | up to 6 months
  Body fat measurements (%)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azabdaftari A, van der Giet M, Schuchardt M, Hennermann JB, Plockinger U, Querfeld U. The cardiovascular phenotype of adult patients with phenylketonuria. Orphanet J Rare Dis. 2019 Sep 6;14(1):213. doi: 10.1186/s13023-019-1188-0. PMID 31492166
- [Background] Berry SA, Brown C, Grant M, Greene CL, Jurecki E, Koch J, Moseley K, Suter R, van Calcar SC, Wiles J, Cederbaum S. Newborn screening 50 years later: access issues faced by adults with PKU. Genet Med. 2013 Aug;15(8):591-9. doi: 10.1038/gim.2013.10. Epub 2013 Mar 7. PMID 23470838
- [Background] Burton BK, Jones KB, Cederbaum S, Rohr F, Waisbren S, Irwin DE, Kim G, Lilienstein J, Alvarez I, Jurecki E, Levy H. Prevalence of comorbid conditions among adult patients diagnosed with phenylketonuria. Mol Genet Metab. 2018 Nov;125(3):228-234. doi: 10.1016/j.ymgme.2018.09.006. Epub 2018 Sep 12. PMID 30266197
- [Background] Cazzorla C, Bensi G, Biasucci G, Leuzzi V, Manti F, Musumeci A, Papadia F, Stoppioni V, Tummolo A, Vendemiale M, Polo G, Burlina A. Living with phenylketonuria in adulthood: The PKU ATTITUDE study. Mol Genet Metab Rep. 2018 Jul 11;16:39-45. doi: 10.1016/j.ymgmr.2018.06.007. eCollection 2018 Sep. PMID 30069431
- [Background] Das AM, Goedecke K, Meyer U, Kanzelmeyer N, Koch S, Illsinger S, Lucke T, Hartmann H, Lange K, Lanfermann H, Hoy L, Ding XQ. Dietary habits and metabolic control in adolescents and young adults with phenylketonuria: self-imposed protein restriction may be harmful. JIMD Rep. 2014;13:149-58. doi: 10.1007/8904_2013_273. Epub 2013 Nov 13. PMID 24222493
- [Background] Ford S, O'Driscoll M, MacDonald A. Living with Phenylketonuria: Lessons from the PKU community. Mol Genet Metab Rep. 2018 Oct 18;17:57-63. doi: 10.1016/j.ymgmr.2018.10.002. eCollection 2018 Dec. PMID 30364670
- [Background] Green B, Browne R, Firman S, Hill M, Rahman Y, Kaalund Hansen K, Adam S, Skeath R, Hallam P, Herlihy I, Jenkinson F, Nicol C, Adams S, Gaff L, Donald S, Dawson C, Robertson L, Fitzachary C, Chan H, Slabbert A, Dunlop C, Cozens A, Newby C, Bittle V, Hubbard G, Stratton R. Nutritional and Metabolic Characteristics of UK Adult Phenylketonuria Patients with Varying Dietary Adherence. Nutrients. 2019 Oct 14;11(10):2459. doi: 10.3390/nu11102459. PMID 31615158
- [Background] Hansen KE, Ney D. A systematic review of bone mineral density and fractures in phenylketonuria. J Inherit Metab Dis. 2014 Nov;37(6):875-80. doi: 10.1007/s10545-014-9735-2. Epub 2014 Jul 9. PMID 25005329
- [Background] Hermida-Ameijeiras A, Crujeiras V, Roca I, Calvo C, Leis R, Couce ML. Arterial stiffness assessment in patients with phenylketonuria. Medicine (Baltimore). 2017 Dec;96(51):e9322. doi: 10.1097/MD.0000000000009322. PMID 29390507
- [Background] MacDonald A, Gokmen-Ozel H, van Rijn M, Burgard P. The reality of dietary compliance in the management of phenylketonuria. J Inherit Metab Dis. 2010 Dec;33(6):665-70. doi: 10.1007/s10545-010-9073-y. Epub 2010 Apr 7. PMID 20373144
- [Background] MacLeod EL, Gleason ST, van Calcar SC, Ney DM. Reassessment of phenylalanine tolerance in adults with phenylketonuria is needed as body mass changes. Mol Genet Metab. 2009 Dec;98(4):331-7. doi: 10.1016/j.ymgme.2009.07.016. Epub 2009 Aug 8. PMID 19747868
- [Background] Okano Y, Hattori T, Fujimoto H, Noi K, Okamoto M, Watanabe T, Watanabe R, Fujii R, Tamaoki T. Nutritional status of patients with phenylketonuria in Japan. Mol Genet Metab Rep. 2016 Aug 20;8:103-10. doi: 10.1016/j.ymgmr.2016.08.005. eCollection 2016 Sep. PMID 27595068
- [Background] Robertson LV, McStravick N, Ripley S, Weetch E, Donald S, Adam S, Micciche A, Boocock S, MacDonald A. Body mass index in adult patients with diet-treated phenylketonuria. J Hum Nutr Diet. 2013 Jul;26 Suppl 1:1-6. doi: 10.1111/jhn.12054. Epub 2013 Apr 3. PMID 23551621
- [Background] Rocha JC, MacDonald A. Dietary intervention in the management of phenylketonuria: current perspectives. Pediatric Health Med Ther. 2016 Dec 1;7:155-163. doi: 10.2147/PHMT.S49329. eCollection 2016. PMID 29388626
- [Background] Rocha JC, MacDonald A, Trefz F. Is overweight an issue in phenylketonuria? Mol Genet Metab. 2013;110 Suppl:S18-24. doi: 10.1016/j.ymgme.2013.08.012. Epub 2013 Aug 31. PMID 24055312
- [Background] Smon A, Groselj U, Zerjav Tansek M, Bicek A, Oblak A, Zupancic M, Krzisnik C, Repic Lampr Et B, Murko S, Hojker S, Battelino T. Newborn Screening in Slovenia. Zdr Varst. 2015 Mar 13;54(2):86-90. doi: 10.1515/sjph-2015-0013. eCollection 2015 Jun. PMID 27646913
- [Background] ten Hoedt AE, de Sonneville LM, Francois B, ter Horst NM, Janssen MC, Rubio-Gozalbo ME, Wijburg FA, Hollak CE, Bosch AM. High phenylalanine levels directly affect mood and sustained attention in adults with phenylketonuria: a randomised, double-blind, placebo-controlled, crossover trial. J Inherit Metab Dis. 2011 Feb;34(1):165-71. doi: 10.1007/s10545-010-9253-9. Epub 2010 Dec 10. PMID 21153445
- [Background] Vockley J, Andersson HC, Antshel KM, Braverman NE, Burton BK, Frazier DM, Mitchell J, Smith WE, Thompson BH, Berry SA; American College of Medical Genetics and Genomics Therapeutics Committee. Phenylalanine hydroxylase deficiency: diagnosis and management guideline. Genet Med. 2014 Feb;16(2):188-200. doi: 10.1038/gim.2013.157. Epub 2013 Oct 10. PMID 24385074
- [Background] van Spronsen FJ, van Wegberg AM, Ahring K, Belanger-Quintana A, Blau N, Bosch AM, Burlina A, Campistol J, Feillet F, Gizewska M, Huijbregts SC, Kearney S, Leuzzi V, Maillot F, Muntau AC, Trefz FK, van Rijn M, Walter JH, MacDonald A. Key European guidelines for the diagnosis and management of patients with phenylketonuria. Lancet Diabetes Endocrinol. 2017 Sep;5(9):743-756. doi: 10.1016/S2213-8587(16)30320-5. Epub 2017 Jan 10. PMID 28082082
- [Background] van Wegberg AMJ, MacDonald A, Ahring K, Belanger-Quintana A, Blau N, Bosch AM, Burlina A, Campistol J, Feillet F, Gizewska M, Huijbregts SC, Kearney S, Leuzzi V, Maillot F, Muntau AC, van Rijn M, Trefz F, Walter JH, van Spronsen FJ. The complete European guidelines on phenylketonuria: diagnosis and treatment. Orphanet J Rare Dis. 2017 Oct 12;12(1):162. doi: 10.1186/s13023-017-0685-2. PMID 29025426
- [Background] Verduci E, Carbone MT, Borghi E, Ottaviano E, Burlina A, Biasucci G. Nutrition, Microbiota and Role of Gut-Brain Axis in Subjects with Phenylketonuria (PKU): A Review. Nutrients. 2020 Oct 29;12(11):3319. doi: 10.3390/nu12113319. PMID 33138040